CLINICAL TRIAL: NCT04774380
Title: A Phase IIIb, Single-arm, Multi-center, International Study of Durvalumab in Combination With Platinum and Etoposide for the First Line Treatment of Patients With Extensive-stage Small Cell Lung Cancer (LUMINANCE)
Brief Title: Study of Durvalumab in Combination With Platinum and Etoposide for the First Line Treatment of Patients With Extensive-stage Small Cell Lung Cancer
Acronym: LUMINANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D419QC00007; 2020-005537-32 (EudraCT Number)
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Extensive-stage Small Cell Lung Cancer
Keywords: Chemotherapy; Aggressive malignancy; Programmed cell death ligand-1; Platinum-based chemotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — durvalumab; Cisplatin; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab - (cisplatin or carboplatin) - Etoposide (Experimental): Participants will receive durvalumab dose A administered via intravenous (IV) infusion concurrently with platinum-based chemotherapy and etoposide every 3 weeks (q3w). Thereafter, durvalumab monotherapy will be continued every 4 weeks post-chemotherapy unless specific treatment discontinuation criteria are met.
  Interventions: Drug: Durvalumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Durvalumab — Participants will receive durvalumab via IV infusion on Day 1 of each cycle.
Drug: Cisplatin — Participants will receive cisplatin via IV administration on Day 1 of each cycle.
Drug: Carboplatin — Participants will receive carboplatin via IV administration Day 1 of each cycle.
Drug: Etoposide — Participants will receive etoposide via IV administration on days 1 to 3 of each cycle.

SUMMARY:
Study to determine the safety and tolerability profile of durvalumab with platinum (cisplatin or carboplatin) plus etoposide (EP) as first-line treatment in participants with extensive-stage small-cell lung cancer.

DETAILED DESCRIPTION:
The study will be conducted in North America, Europe and Turkey.

In this single arm study participants will be treated with with durvalumab alone and concurrently with platinum-based chemotherapy and etoposide during the study period until radiological disease progression, unless there is clinical progression, unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met, as per investigator assessment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-documented ES-SCLC (stage IV [T any, N any, M1 a/b], or with T3-4 due to multiple lung nodules that are too extensive or have tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan (Brain metastases; must be asymptomatic or treated and stable off steroids and anticonvulsants for at least 1 month prior to study treatment)
* Participants must be considered suitable to receive a platinum-based chemotherapy regimen as 1st line treatment for the ES-SCLC. Chemotherapy must contain either cisplatin or carboplatin in combination with etoposide
* World Health Organization/ Eastern Cooperative Oncology Group performance status of 0 to 2 at enrollment Baseline computed tomography/ magnetic resonance imaging results of the brain, chest and abdomen (including liver and adrenal glands) within 28 days prior to the treatment initiation
* No prior exposure to immune-mediated therapy including, but not limited to, other anti- CTLA-4, anti-Programmed cell death-1 (PD-1), anti- Programmed cell death ligand-1 (PD-L1), and anti-PD-L2 (anti-PD-L2) antibodies, excluding therapeutic anticancer vaccines
* Adequate organ and marrow function
* Body weight > 30 kg
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal participants

Exclusion Criteria:

* History of allogeneic organ transplantation
* Active or prior documented autoimmune or inflammatory disorders, systemic lupus erythematosus, sarcoidosis syndrome, or wegener syndrome
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, active interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the participant to give written informed consent
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease ≥ 5 years before the first dose of Investigational medicinal product (IMP) and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* History of leptomeningeal carcinomatosis and active primary immunodeficiency
* Active infection including tuberculosis, hepatitis B, hepatitis C, human immunodeficiency virus
* Any unresolved toxicity Common Terminology Criteria for Adverse Events Grade ≥ 2 from previous anticancer therapy
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
* Received prior systemic therapy for ES-SCLC
* Medical contraindication to platinum (cisplatin or carboplatin)-etoposide-based chemotherapy
* Any concurrent chemotherapy, IMP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions is acceptable
* Planned consolidation chest radiation therapy. Radiation therapy outside of the chest for palliative care is allowed but must be completed before first dose of the study medication
* Receipt of live attenuated vaccine within 30 days prior to the first dose of in IMP
* Major surgical procedure within 28 days prior to the first dose of IMP
* Participants who have received prior immunotherapy agents including anti-PD-1 or anti PD-L1
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab
* Participation in another clinical study with an investigational product administered in the last 4 weeks
* Female participants who are pregnant or breastfeeding or male or female participants of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab and 180 days after the last dose of etoposide

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2025-01-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- Bulgaria (3):
  - Research Site, Panagyurishte
  - Research Site, Rousse
  - Research Site, Sofia
- Research Site, Montreal, Quebec, Canada
- Czechia (3):
  - Research Site, Burgas
  - Research Site, Olomouc
  - Research Site, Ostrava
- Germany (6):
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Gauting
  - Research Site, Hamburg
  - Research Site, Jena
  - Research Site, Kassel
- Italy (7):
  - Research Site, Ancona
  - Research Site, Bari
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Orbassano
  - Research Site, Palermo
  - Research Site, Roma
- Turkey (Türkiye) (9):
  - Research Site, Adapazarı
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Bursa
  - Research Site, Edirne
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Malatya
  - Research Site, Pamukkale

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419QC00007&attachmentIdentifier=63ae71a0-e925-417e-ad33-008bce95d9c5&fileName=D419QC00007_Redacted_CSP.pdf&versionIdentifier=
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419QC00007&attachmentIdentifier=224e7482-7a07-4739-ad7b-c78d01bc5f72&fileName=D419QC00007_Redacted_CSR_synopsis.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419QC00007&attachmentIdentifier=447ccb65-152f-4e82-8bb4-7a2f151dfdb3&fileName=D419QC00007_Redacted_SAP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 32 sites in 5 countries: Bulgaria, Czech Republic, Germany, Italy, Turkey. Study results are presented as of final data cut-off (DCO), 21Apr2024. After final DCO, no additional data was collected for the purpose of the analysis. Participants were allowed to continue the study drug until other drug supply options were available. The last subject's last visit was declared on 2Jan2025 once all participants were transferred to a rollover study or marketed product.
Pre-assignment Details: Participants who met all the inclusion and none of the exclusion criteria were enrolled in this study. All study assessments were performed as per the schedule of assessment.
Groups:
- Durvalumab - (Cisplatin or Carboplatin) - Etoposide (Durvalumab +EP): Participants received durvalumab 1500 mg administered via intravenous (IV) infusion concurrently with platinum-based chemotherapy and etoposide every 3 weeks (q3w) up to 6 cycles. Thereafter, durvalumab monotherapy was continued every 4 weeks post-chemotherapy unless specific treatment discontinuation criteria were met.
Period: Overall Study
Arm/Group | Durvalumab - (Cisplatin or Carboplatin) - Etoposide (Durvalumab +EP)
Started | 152
Completed (Patients who terminated study) | 152 (44 patients were ongoing study at final DCO.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF) which consisted of all enrolled patients who received at least 1 dose of any study treatment.
Groups:
- Durvalumab +EP: Participants received durvalumab 1500 mg administered IV infusion concurrently with platinum-based chemotherapy and etoposide every 3 weeks (q3w) up to 6 cycles. Thereafter, durvalumab monotherapy was continued every 4 weeks post-chemotherapy unless specific treatment discontinuation criteria were met.
Arm/Group | Durvalumab +EP
Number analyzed (Participants) | 152
Age, Continuous [Median (Full Range); unit: Years] | 64.0 [27 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 98
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 151
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incidence of Grade 3 or Higher Adverse Events (AEs)
Description: Incidence of Grade 3 or higher adverse events to evaluate safety and tolerability profile of durvalumab + Platinum (cisplatin or carboplatin) plus etoposide (EP) treatment was assessed.
Time Frame: From first dose of study treatment until 90 days after treatment discontinuation, up to 2.5 years.
Population: SAF which consisted of all enrolled patients who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Durvalumab+EP: Participants received durvalumab 1500 mg via IV infusion concurrently with platinum-based chemotherapy and etoposide every 3 weeks (q3w) up to 6 weeks. Thereafter, durvalumab monotherapy was continued every 4 weeks post-chemotherapy unless specific treatment discontinuation criteria were met.
Arm/Group | Durvalumab+EP
Number analyzed (Participants) | 152
Participants | 91

2. Primary Outcome: Number of Participants With Incidence of Immune Mediated Adverse Events (imAEs)
Description: Immune mediated adverse events (imAEs) were assessed to evaluate safety and tolerability profile of durvalumab + EP treatment. An imAE is defined as an AESI that is associated with drug exposure and is consistent with an immune-mediated mechanism of action (MOA) and where there is no clear alternate etiology.
Time Frame: From first dose of study treatment until 90 days after treatment discontinuation, up to 2.5 years.
Population: SAF which consisted of all enrolled patients who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab+EP
Number analyzed (Participants) | 152
Participants | 22

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Efficacy of durvalumab + EP treatment by evaluating PFS according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) was assessed. The PFS is the time from the first date of treatment until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the participant withdrew from Investigational medicinal product (IMP) or received another anticancer therapy prior to progression.
Time Frame: From first dose of study treatment until disease progression or death, up to 2.5 years.
Population: SAF which consisted of all enrolled patients who received at least 1 dose of any study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab+EP
Number analyzed (Participants) | 152
Months | 6.3 [5.75 to 6.47]

4. Secondary Outcome: Percentage of Participants Alive and Progression-free at 12 Months From First Date of Treatment (PFS12)
Description: The efficacy of durvalumab + EP treatment by evaluating PFS12 according to RECIST 1.1 was assessed.
Time Frame: From first date of study treatment until 12 months.
Population: SAF which consisted of all enrolled patients who received at least 1 dose of any study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Durvalumab+EP
Number analyzed (Participants) | 152
Percentage of participants | 15.0 [9.76 to 21.21]

5. Secondary Outcome: Objective Response Rate (ORR)
Description: The efficacy of durvalumab + EP treatment by evaluating ORR according to RECIST 1.1 was assessed. The ORR will be assessed based on Investigator-assessed response to treatment of complete response (CR) and partial response (PR), per RECIST1.1.
Time Frame: From screening until disease progression or the last evaluable assessment in the absence of progression, up to 2.5 years.
Population: SAF which consisted of all enrolled patients who received at least 1 dose of any study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Durvalumab+EP
Number analyzed (Participants) | 152
Percentage of participants | 66.4 [58.3 to 73.9]

6. Secondary Outcome: Duration of Response (DoR)
Description: The efficacy of durvalumab + EP treatment by evaluating DoR according to RECIST 1.1 was assessed. The DoR is time from the date of first documented response per RECIST1.1 until the first date of documented progression per RECIST1.1 or death in the absence of disease progression.
Time Frame: From the date of first documented response until the first date of documented progression or death in the absence of disease progression, up to 2.5 years.
Population: SAF which consisted of all enrolled patients who received at least 1 dose of any study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab+EP
Number analyzed (Participants) | 101
Months | 5.2 [5.03 to 5.59]

7. Secondary Outcome: Percentage of Participants Remaining in Response, 12 Months After First Documented Objective Response (DoR12)
Description: The efficacy of durvalumab + EP treatment by evaluating DoR12 according to RECIST 1.1 was assessed.
Time Frame: as for outcome 6
Population: SAF which consisted of all enrolled patients who received at least 1 dose of any study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Durvalumab+EP
Number analyzed (Participants) | 101
Percentage of participants | 19.8 [12.70 to 28.06]

8. Secondary Outcome: Overall Survival (OS)
Description: Assessment of the efficacy of durvalumab + EP treatment by evaluating OS. The OS is the time from the first date of treatment until death due to any cause.
Time Frame: From first dose of study treatment to death, up to 2.5 years.
Population: SAF which consisted of all enrolled patients who received at least 1 dose of any study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab+EP
Number analyzed (Participants) | 152
Months | 16.4 [12.45 to 18.73]

9. Secondary Outcome: Percentage of Participants Alive at 12 Months From First Date of Treatment (OS12)
Description: The efficacy of durvalumab + EP treatment by evaluating OS12 was assessed.
Time Frame: From first dose of study treatment till 12 months.
Population: SAF which consisted of all enrolled patients who received at least 1 dose of any study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Durvalumab+EP
Number analyzed (Participants) | 152
Percentage of participants | 59.8 [51.00 to 67.55]

10. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: To evaluate safety and tolerability profile of durvalumab + EP treatment, adverse events and serious adverse events were assessed.
Time Frame: From first dose of study treatment until 90 days after discontinuation, up to 2.5 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab+EP
Number analyzed (Participants) | 152
Participants
  Any Adverse event (AE) | 142
  Any AE possibly related to any treatment | 109
  Any AE of maximum CTCAE grade 3 or grade 4 | 85
  Any AE of maximum CTCAE grade 3 or grade 4, possibly related to any treatment | 59
  Any AE with outcome of death | 15
  Any AE with outcome of death, possibly related to any treatment | 4
  Any AE with outcome of death, possibly related to durvalumab | 0
  Any AE with outcome of death, possibly related to EP | 4
  Any SAE (including events with outcome of death) | 52
  Any SAE (including events with outcome of death), possibly related to any treatment | 16
  Any AE leading to interruption or discontinuation of durvalumab | 40
  Any AE leading to interruption or discontinuation of EP | 41

11. Secondary Outcome: Number of Participants With Adverse Events of Special Interests
Description: To evaluate safety and tolerability profile of durvalumab + EP treatment, adverse events of special interests were assessed. An AESI is an AE of scientific and medical interest specific to understanding of the IMP. AESIs for durvalumab include, but are not limited to, events with a potential inflammatory or immune-mediated mechanism and which may require more frequent monitoring and/or interventions such as steroids, immunosuppressants, and/or hormone replacement therapy.
  This includes adverse events of special/ possible interest.
Time Frame: From first dose of study treatment until 90 days after discontinuation, up to 2.5 years.
Population: SAF which consisted of all enrolled patients who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab+EP
Number analyzed (Participants) | 152
Participants | 82

ADVERSE EVENTS:
Time Frame: From first dose of study treatment until 90 days after treatment discontinuation, up to 2.5 years.
Arm/Group | Durvalumab+EP
All-Cause Mortality (participants affected / at risk) | 85/152
Serious Adverse Events (participants affected / at risk) | 52/152
Other Adverse Events (participants affected / at risk) | 136/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab+EP (N=152)
Abdominal infection (Infections and infestations) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 9 (9)
Postoperative wound infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Tooth abscess (Infections and infestations) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4)
Brain oedema (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Embolism arterial (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (2)
Superior vena cava syndrome (Vascular disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Cellulite (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (5)
Death (General disorders) | 1 (1)
Swelling (General disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 3 (3)
Urine output decreased (Investigations) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Immune-mediated encephalopathy (Nervous system disorders) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Suspected drug-induced liver injury (Hepatobiliary disorders) | 1 (1)
Intestinal anastomosis (Surgical and medical procedures) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.03% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab+EP (N=152)
COVID-19 (Infections and infestations) | 10 (10)
Upper respiratory tract infection (Infections and infestations) | 13 (16)
Anaemia (Blood and lymphatic system disorders) | 85 (117)
Leukocytosis (Blood and lymphatic system disorders) | 7 (8)
Leukopenia (Blood and lymphatic system disorders) | 19 (30)
Neutropenia (Blood and lymphatic system disorders) | 51 (91)
Thrombocytopenia (Blood and lymphatic system disorders) | 24 (44)
Hyperthyroidism (Endocrine disorders) | 18 (28)
Hypothyroidism (Endocrine disorders) | 18 (22)
Decreased appetite (Metabolism and nutrition disorders) | 13 (13)
Hypermagnesaemia (Metabolism and nutrition disorders) | 5 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 (13)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 19 (24)
Hyponatraemia (Metabolism and nutrition disorders) | 15 (21)
Dizziness (Nervous system disorders) | 8 (8)
Headache (Nervous system disorders) | 11 (13)
Neuropathy peripheral (Nervous system disorders) | 6 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (7)
Hypotension (Vascular disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (13)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 7 (8)
Constipation (Gastrointestinal disorders) | 30 (35)
Diarrhoea (Gastrointestinal disorders) | 13 (18)
Dyspepsia (Gastrointestinal disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 37 (56)
Stomatitis (Gastrointestinal disorders) | 8 (9)
Vomiting (Gastrointestinal disorders) | 8 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 20 (20)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6)
Asthenia (General disorders) | 10 (11)
Fatigue (General disorders) | 24 (29)
Oedema peripheral (General disorders) | 6 (7)
Pyrexia (General disorders) | 12 (13)
Alanine aminotransferase increased (Investigations) | 12 (14)
Amylase increased (Investigations) | 9 (9)
Aspartate aminotransferase increased (Investigations) | 14 (18)
Blood alkaline phosphatase increased (Investigations) | 10 (13)
Blood creatinine increased (Investigations) | 18 (25)
Blood lactate dehydrogenase increased (Investigations) | 9 (10)
Gamma-glutamyltransferase increased (Investigations) | 15 (17)
Lipase increased (Investigations) | 6 (6)
Neutrophil count decreased (Investigations) | 15 (24)
Platelet count decreased (Investigations) | 12 (19)
Weight decreased (Investigations) | 8 (9)
White blood cell count decreased (Investigations) | 16 (25)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (6)
Dermatitis (Skin and subcutaneous tissue disorders) | 5 (6)
Depression (Psychiatric disorders) | 5 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 5 (6)

LIMITATIONS AND CAVEATS:
The study results are presented as of the final data cut-off dated April 21, 2024. After final DCO, no additional data was collected for the purpose of the analysis. The participants were allowed to continue the study drug until other drug supply options were available. The last subject's last visit was declared once all participants were transferred to a rollover study or a marketed product, which occurred on January 2, 2025 and was reported as the study completion date.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2021-08-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT04774380/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT04774380/SAP_001.pdf